CLINICAL TRIAL: NCT01508858
Title: A Double-blind, Two Period Cross-over, Single Centre Trial in Healthy Subjects Investigating the Influence on the Pharmacokinetics of Ethinylestradiol and Levonorgestrel in an Oral Contraceptive Drug After Multiple Dose Administration of Liraglutide
Brief Title: Influence on the Effect of an Oral Contraceptive Drug After Administration of Liraglutide in Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1330; 2006-003904-21 (EudraCT Number)
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Levonorgestrel; Ethinyl Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment period 1 (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo; Drug: levonorgestrel / ethinylestradiol
- Treatment period 2 (Placebo Comparator)
  Interventions: Drug: liraglutide; Drug: placebo; Drug: levonorgestrel / ethinylestradiol

INTERVENTIONS:
Drug: liraglutide — Administered with daily subcutaneous injections for approximately 3 weeks in each treatment period in random order
Drug: placebo — Administered with daily subcutaneous injections for approximately 3 weeks in each treatment period in random order
Drug: levonorgestrel / ethinylestradiol — One single oral tablet after the liraglutide or placebo dose administration at the end of each treatment period

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate if liraglutide changes AUC (area under the curve) of ethinylestradiol and levonorgestrel administered as a combination contraceptive drug (Neovletta®).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal woman
* Body Mass Index (BMI) between 18.0-30.0 kg/m^2 (both inclusive)
* Good general health as judged by the investigator, based on medical history, physical examination including 12-lead ECG (electrocardiogram), vital signs, blood and urinary laboratory assessments

Exclusion Criteria:

* History of any clinically significant renal, hepatic, cardiovascular, pulmonary, gastrointestinal, metabolic, endocrine, haematological, neurological, psychiatric disease or other major disorders that may interfere with the objectives of the trial, as judged by the investigator
* Impaired renal function
* Active hepatitis B and/or active hepatitis C
* Positive HIV (human immunodeficiency virus) antibodies
* Known or suspected allergy to trial products or related products
* Pregnant or positive pregnancy test at screening or nursing mother
* Use of prescription or non-prescription medication within 2 weeks prior to first dosing with trial products which in the Investigators opinion will interfere with the pharmacokinetics of the compounds in Neovletta®
* Use of hormone replacement therapy within 4 weeks prior to starting dosing with trial product
* History of alcoholism or drug abuse
* Smoking of more than 10 cigarettes per day, or the equivalent for other tobacco products
* Habitual excessive consumption of methylxanthine-containing beverages and foods (coffee, tea, soft drinks such as cola, chocolate) as judged by the Investigator
* Excessive consumption of a diet deviating from a normal diet as judged by the Investigator

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
AUC of ethinylestradiol
AUC of levonorgestrel

SECONDARY OUTCOMES:
AUC (0-t)
Cmax, maximum concentration
tmax, time to reach Cmax
t½, terminal half-life
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Uppsala, Sweden

REFERENCES:
- [Result] Jensen TM, Saha K, Steinberg WM. Is there a link between liraglutide and pancreatitis? A post hoc review of pooled and patient-level data from completed liraglutide type 2 diabetes clinical trials. Diabetes Care. 2015 Jun;38(6):1058-66. doi: 10.2337/dc13-1210. Epub 2014 Dec 12. PMID 25504028
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com